CLINICAL TRIAL: NCT07025902
Title: Holistic Support Pathways for Maternal Psychological Wellbeing: A Comprehensive Approach From Preconception to Postpartum (SOS-Mamma).
Brief Title: Screening for Postpartum Depression Using EPDS and HAM-D in Mothers Within 72 Hours After Delivery at a Tertiary Care Center (SOS-Mamma Study)
Acronym: SOS-Mamma
Status: Not yet recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Marco La Verde, M.D., researcher and PhD student, University of Campania Luigi Vanvitelli
Other Study IDs: 0017100/i
Record Dates: First submitted 2025-06-09; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Post Partum Depression
Keywords: Post Partum Depression; EPDS; HAM-D Scales
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postpartum Women Screened Within 72 Hours After Delivery: This cohort consists of postpartum women who deliver a live-born infant at ≥35 weeks of gestation and are clinically stable. Participants are screened within 72 hours after childbirth using the Edinburgh Postnatal Depression Scale (EPDS) and the Hamilton Depression Rating Scale (HAM-D). The study includes both women with and without depressive symptoms, allowing comparison within the cohort based on screening results. The purpose is to assess the incidence of postpartum depression and identify associated socio-demographic or obstetric risk factors in a real-world clinical setting
  Interventions: Diagnostic Test: Standardized Psychological Screening Using EPDS and HAM-D

INTERVENTIONS:
Diagnostic Test: Standardized Psychological Screening Using EPDS and HAM-D — Participants will undergo a standardized psychological screening protocol for postpartum depression within 72 hours after delivery. The protocol includes: (1) completion of the Edinburgh Postnatal Depression Scale (EPDS), a 10-item self-administered questionnaire assessing depressive symptoms; and (2) administration of the Hamilton Depression Rating Scale (HAM-D), a 17-item clinician-administered tool for evaluating the severity of depressive symptoms. The combined use of these tools allows early detection and stratification of postpartum depressive symptoms in a clinical population.

SUMMARY:
Postpartum depression (PPD) is one of the most common complications affecting maternal mental health after childbirth, with an estimated prevalence of 10-20% in high-income countries. Despite its frequency and the availability of effective screening tools, early diagnosis remains largely underestimated in routine clinical care.

This study, part of the national SOS-Mamma project funded by the Italian Ministry of Health, aims to systematically screen for signs of postpartum depression in women giving birth at a tertiary care obstetric unit (AOU Vanvitelli - UOC of Obstetrics and Gynecology, Naples, Italy). The goal is to promote early detection and timely referral to specialized care pathways.

The study is a prospective, observational, monocentric, non-interventional, non-pharmacological study. All eligible women who deliver at the hospital will be invited to participate within the first 72 hours after childbirth. Participants will be asked to complete the Edinburgh Postnatal Depression Scale (EPDS) - a widely used self-report questionnaire - and will undergo a brief clinical interview using the Hamilton Depression Rating Scale (HAM-D), conducted by trained healthcare staff.

The study's primary objective is to estimate the real-world incidence of postpartum depression within this population. Secondary objectives include identifying socio-demographic and obstetric risk factors associated with depressive symptoms, assessing the acceptability and feasibility of routine screening, and contributing to the development of a replicable model of care aligned with international recommendations (NICE, WHO, ISS).

Collected data will be anonymized and analyzed to provide evidence on early indicators of PPD and guide improvements in clinical care. Women identified as being at risk (e.g., EPDS >10 or presence of suicidal ideation) will be referred to specialist psychiatric services in accordance with clinical guidelines.

Participation in the study is voluntary. All procedures comply with European data protection regulations and Good Clinical Practice (GCP) principles. No experimental treatments are involved, and no changes to standard care will be made based on study participation.

By highlighting the need for structured mental health screening in the postpartum period, this study hopes to improve maternal wellbeing and reduce the long-term impact of undiagnosed depression on mothers and their children.

DETAILED DESCRIPTION:
This clinical study is part of the national project SOS-Mamma ("Holistic Support Pathways for Maternal Psychological Wellbeing"), funded by the Italian Ministry of Health (Programma CCM 2024). The present protocol outlines a prospective, observational, monocentric, non-pharmacological, non-interventional study, aiming to estimate the incidence of postpartum depression (PPD) and evaluate the clinical feasibility of implementing a standardized screening protocol in a real-life maternity care setting.

The study is conducted at a tertiary-level obstetric and gynecologic unit (AOU Vanvitelli - UOC of Obstetrics and Gynecology, Naples, Italy), over a planned recruitment period of 24 months. Eligible participants include women delivering live-born infants at ≥35 weeks of gestation, who are clinically stable, able to consent, and able to complete the questionnaires in Italian or English.

Screening Protocol

Within 72 hours after delivery, enrolled participants will undergo a standardized two-step screening process for depressive symptoms:

Edinburgh Postnatal Depression Scale (EPDS): a validated self-administered questionnaire assessing depressive symptoms over the previous two weeks.

Hamilton Depression Rating Scale (HAM-D): a clinician-administered scale evaluating the severity of depressive symptoms via a 17-item structured interview.

Clinical, socio-demographic, and obstetric data will be collected from medical records and patient interviews, including maternal age, parity, education level, marital status, occupational status, pregnancy complications, delivery mode, neonatal outcomes (e.g., Apgar score, NICU admission), and psychiatric history.

Primary Objective To estimate the incidence of postpartum depression within 72 hours postpartum using validated screening instruments (EPDS and HAM-D) in a real-world clinical population.

Secondary Objectives To identify clinical and socio-demographic risk factors associated with depressive symptoms.

To assess the feasibility and acceptability of implementing a systematic screening protocol in postpartum care.

To generate evidence for a scalable model of early detection and referral for maternal mental health disorders in accordance with international guidelines (NICE, WHO, ISS).

Sample Size and Statistical Considerations Based on previous epidemiological data (expected prevalence of PPD ~19% in the local population), a sample size of at least 273 women is calculated to detect ≥53 cases of postpartum depression, with an alpha of 0.05 and statistical power >80%. This sample will allow for robust estimation of incidence and risk factor associations.

Data analysis will include descriptive statistics, bivariate comparisons (e.g., chi-square test, t-test, Mann-Whitney U), and multivariate logistic regression models to identify independent predictors of depressive symptoms. The software MedCalc (v23.2.1) will be used for all analyses.

Quality Assurance and Data Management Data anonymization will be implemented immediately after collection using a study-specific alphanumeric code.

Data will be stored in a secure, password-protected electronic database accessible only to authorized research personnel.

Data quality control will include double entry checks, logic checks for consistency and range, and periodic review by the Principal Investigator.

The study team will follow Standard Operating Procedures (SOPs) for recruitment, informed consent, questionnaire administration, data recording, and adverse event documentation.

All research staff involved in data collection and screening will be trained in Good Clinical Practice (GCP) and use of the screening instruments.

Adverse events (including psychological distress triggered by the screening process) will be recorded, reported, and referred to psychiatric evaluation per protocol.

Handling of Missing Data In case of missing, inconsistent, or uninterpretable data, predefined coding will be used to distinguish between non-response, refusal, technical error, or medical unsuitability. Missing data will be analyzed descriptively and handled via appropriate imputation or exclusion methods depending on their frequency and pattern.

Ethical and Regulatory Compliance This study will be conducted in accordance with the Declaration of Helsinki, GCP, GDPR (EU Regulation 2016/679), and applicable national laws. Ethical approval has been requested from the competent ethics committee, and informed consent will be obtained from all participants.

Dissemination and Transparency Findings will be submitted for peer-reviewed publication and presented at scientific conferences, irrespective of the outcome. The dataset may be made available for secondary analysis upon justified request, following ethical and regulatory approval.

ELIGIBILITY:
nclusion Criteria

Women aged ≥18 and <45 years at the time of delivery

Singleton pregnancy at term (≥37 weeks) or late preterm (≥35 weeks of gestation)

Live-born infant in clinically stable condition at discharge

Ability to understand and complete self-reported questionnaires (EPDS) in Italian or English

Ability to provide written informed consent

Screening performed within 72 hours postpartum during routine hospital stay

Exclusion Criteria

Multiple pregnancy (e.g., twins or higher-order gestations)

Major psychiatric diagnosis under active treatment at the time of delivery (e.g., schizophrenia, bipolar disorder)

Severe language barriers preventing adequate understanding of the consent form or questionnaires

Neonatal death or congenital anomalies requiring prolonged NICU admission

Maternal age <18 or ≥45 years at delivery

Gestational age at birth <35 weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is restricted to biological females who have recently delivered a live-born infant. The study targets postpartum women within 72 hours after childbirth in order to assess early depressive symptoms related to the perinatal period. Individuals identifying as women but not having given birth are not eligible. Gender-based eligibility is therefore directly related to the biological and clinical characteristics of postpartum status, which is central to the study objectives.
Study Population: The study population consists of postpartum women who deliver at the AOU Vanvitelli - UOC of Obstetrics and Gynecology, a tertiary care academic hospital in Naples, Italy. This is a real-world clinical population composed primarily of women receiving routine obstetric care through the Italian National Health System. The cohort includes patients with both physiological and low-risk obstetric complications. Participants will be recruited during their standard postpartum hospital stay, within 72 hours after delivery.
Sampling Method: Probability Sample
Enrollment: 273 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postpartum depression assessed by EPDS | Within 72 hours postpartum during routine hospital stay following delivery
  Incidence of postpartum depression assessed by EPDS The proportion of postpartum women who screen positive for depressive symptoms within 72 hours after delivery, based on the Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a 10-item self-report questionnaire, and a score ≥10 is considered indicative of clinically relevant depressive symptoms.
Incidence of postpartum depression assessed by HAM-D | Within 72 hours postpartum during routine hospital stay following delivery
  The proportion of postpartum women who screen positive for depressive symptoms within 72 hours after delivery, based on the Hamilton Depression Rating Scale (HAM-D). This clinician-administered scale assesses severity of depression; established cutoff scores will be used to classify presence of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Largo Madonna delle grazie 1, Naples, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers. The informed consent form signed by participants does not include provisions for data sharing outside the study team. Additionally, due to the sensitive nature of mental health data and the single-site observational design, sharing of IPD is not planned in order to ensure full compliance with ethical and data protection regulations (including GDPR).

REFERENCES:
- [Result] Luciano M, Di Vincenzo M, Brandi C, Tretola L, Toricco R, Perris F, Volpicelli A, Torella M, La Verde M, Fiorillo A, Sampogna G. Does antenatal depression predict post-partum depression and obstetric complications? Results from a longitudinal, long-term, real-world study. Front Psychiatry. 2022 Dec 14;13:1082762. doi: 10.3389/fpsyt.2022.1082762. eCollection 2022. PMID 36590632